CLINICAL TRIAL: NCT07325656
Title: Comparison of Scoring Systems for Predicting Morbidity and Mortality in Patients Undergoing Surgery for Gastrointestinal Malignancies
Brief Title: Comparison of Scoring Systems in Gastrointestinal Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Lütfi Kırdar City Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Emre Gecici, Specialist Physician, Lütfi Kırdar City Hospital
Other Study IDs: LutfiKırdarCityHospital
Record Dates: First submitted 2025-11-30; First posted 2026-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastro Intestinal Cancer; Scoring Systems
Keywords: mortality; morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastrointestinal Cancer Surgery Cohort: Prospective observational group including adult patients undergoing elective surgery for gastrointestinal malignancy. Risk prediction scores will be recorded pre- and peri-operatively.

SUMMARY:
Accurate prediction of postoperative morbidity and mortality is essential for optimizing perioperative management in patients undergoing gastrointestinal cancer surgery. This study evaluates the predictive performance of commonly used perioperative risk scoring systems in patients undergoing gastrointestinal surgery for malignancy under general anesthesia.

DETAILED DESCRIPTION:
This prospective observational study is designed to assess the predictive accuracy of multiple perioperative risk assessment tools in adult patients undergoing gastrointestinal (GI) surgery for malignancy under general anesthesia. Preoperative risk stratification is a key component of perioperative care, as it supports identification of patients at increased risk for postoperative complications and mortality and facilitates appropriate perioperative planning and resource utilization.

Perioperative risk scores are calculated using routinely collected clinical data obtained during the preoperative evaluation and intraoperative period, in accordance with established definitions for each scoring system. The scoring systems evaluated include the American Society of Anesthesiologists Physical Status classification (ASA-PS), Surgical Apgar Score (SAS), Portsmouth Physiological and Operative Severity Score for the Enumeration of Mortality and Morbidity (P-POSSUM), American College of Surgeons National Surgical Quality Improvement Program Surgical Risk Calculator (ACS-NSQIP-SRC), and the ARISCAT risk score for postoperative pulmonary complications.

Postoperative outcomes are assessed during the index hospitalization and early postoperative follow-up period, focusing on the occurrence of pulmonary and non-pulmonary complications, short-term mortality, requirement for intensive care unit admission, and length of hospital and intensive care unit stay.

The primary objective of the study is to determine which perioperative risk assessment tools demonstrate the highest predictive accuracy for postoperative complications and mortality following gastrointestinal malignancy surgery. Secondary objectives include comparison of score performance for pulmonary versus non-pulmonary complications and evaluation of associations between risk scores and postoperative length of stay.

The results of this study are expected to provide clinically relevant evidence regarding the utility of commonly used perioperative risk scoring systems in gastrointestinal cancer surgery and to support improved perioperative risk stratification.

ELIGIBILITY:
Inclusion Criteria: Age ≥ 18 years, Scheduled to undergo elective gastrointestinal surgery for malignancy via laparotomy, Planned general anesthesia, Provision of written informed consent

Exclusion Criteria: Emergency surgery, Surgery performed using laparoscopic or robotic approaches, Previous gastrointestinal surgery for malignancy within the past 6 months, Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (≥18 years) scheduled for elective gastrointestinal malignancy surgery performed under general anesthesia at a tertiary referral hospital. Participants are followed prospectively from the preoperative assessment through the postoperative period. Demographic characteristics, baseline clinical data, and operative variables are collected. Postoperative clinical outcomes are assessed to evaluate the predictive performance of perioperative risk scoring systems for postoperative morbidity and mortality.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
30- and 60-day All-Cause Postoperative Mortality | 60 days after surgery
  All-cause mortality within 30 and 60 days after gastrointestinal malignancy surgery performed under general anesthesia. Mortality data will be obtained from hospital records and verified through national health databases.

SECONDARY OUTCOMES:
Postoperative Pulmonary Complications | Within 30 days after surgery
  Occurrence of any pulmonary complication including pneumonia, respiratory failure requiring reintubation or mechanical ventilation >24 hours, bronchospasm, pulmonary edema, or atelectasis as defined by ARISCAT/EPCO criteria.

OTHER OUTCOMES:
Postoperative Non-Pulmonary Complications | Within 30 days after surgery
  Occurrence of any non-pulmonary postoperative complication such as wound infection, sepsis, acute kidney injury, postoperative bleeding, cardiac event (arrhythmia, myocardial infarction, heart failure), or ileus.

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET E GECICI, MD, Principal Investigator — Kartal Dr. Lutfi Kirdar City Hospital
Locations (1):
- Kartal Dr. Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vashistha N, Singhal S, Budhiraja S, Singhal D. Evaluation of ACS-NSQIP and CR-POSSUM risk calculators for the prediction of mortality after colorectal surgery: A retrospective cohort study. J Minim Access Surg. 2024 Apr 1;20(2):142-147. doi: 10.4103/jmas.jmas_187_22. Epub 2022 Sep 12. PMID 36124474
- [Result] Nag DS, Dembla A, Mahanty PR, Kant S, Chatterjee A, Samaddar DP, Chugh P. Comparative analysis of APACHE-II and P-POSSUM scoring systems in predicting postoperative mortality in patients undergoing emergency laparotomy. World J Clin Cases. 2019 Aug 26;7(16):2227-2237. doi: 10.12998/wjcc.v7.i16.2227. PMID 31531317
- [Result] Crea N, Di Fabio F, Pata G, Nascimbeni R. APACHE II, POSSUM, and ASA scores and the risk of perioperative complications in patients with colorectal disease. Ann Ital Chir. 2009 May-Jun;80(3):177-81. PMID 20131533

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT07325656/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT07325656/ICF_001.pdf